CLINICAL TRIAL: NCT02450123
Title: Single-arm Study to Evaluate the Safety and Efficacy of Sunitinib, in Subjects With RET Fusion Positive or FGFR2 Amplification, Refractory Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-076
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sunitinib (Experimental): sunitinib 50mg will be administered orally once a day 42 days.Study treatment will be continued until objective disease progression.
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib
  Other Names: sutene

SUMMARY:
This is a pilot study of sunitinib in patients with RET fusion positive or FGFR2 Amplification Refractory solid tumors.

This study is a single-arm, pilot study of sunitinib in subjects with Refractory solid tumors harboring RET fusion positive or FGFR2 Amplification sunitinib 50mg will be administered orally once a day 42 days.Study treatment will be continued until objective disease progression.

To investigate the efficacy of sunitinib in subjects with Refractory solid tumors harboring RET fusion positive or FGFR2 Amplification.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. RET fusion positive,FGFR amplification, Refractory Solid Tumors that has recurred or progressed following standard therapy, or that has not responded to standard therapy, or for which there is no standard therapy.
4. ECOG performance status 0-2.
5. Have measurable or evaluated disease based on RECIST1.1. as determined by investigator.
6. Adequate Organ Function Laboratory Values

   * Absolute neutrophil count ≥ 1.5 x 109/L, Hemoglobin ≥ 9g/dL, Platelets ≥ 75 x 109/L
   * bilirubin ≤ 1.5 x upper limit of normal AST/ALT ≤ 2.5 x upper limit of normal (5.0 X upper limit of normal , for subjects with liver metastases)
   * creatinine ≤1.5 x UNL
7. Patients of child-bearing potential should be using adequate contraceptive measures (two forms of highly reliable methods) should not be breast feeding and must have a negative pregnancy test prior to start of dosing.
8. Adequate heart function.

Exclusion Criteria:

1. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
2. Has known active central nervous system (CNS) metastases.
3. Has an active infection requiring systemic therapy.
4. Pregnancy or breast feeding
5. Patients with cardiac problem.
6. Any previous treatment with sunitinib

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
progression-free survival | expected average of 24 weeks

SECONDARY OUTCOMES:
objective response rate | expected average of 24 weeks
Time to progression | expected average of 24 weeks
overall survival | expected average of 24 weeks
Number of subjects with Adverse Events as a measure of toxicity profile | expected average of 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea